CLINICAL TRIAL: NCT05408806
Title: The Effect of Technology Assisted Rehabilitation Interventions on Postural Control, Activity and Participation in Children With Cerebral Palsy
Brief Title: Technology Assisted Rehabilitation in CP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Yonca Zenginler Yazgan, Asst. Prof., Istanbul University - Cerrahpasa
Other Study IDs: E-74555795-050.01.04-346301
Record Dates: First submitted 2022-05-25; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; postural control; rehabilitation; virtual reality games; hippotherapy simulator
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Virtual Reality Games Group with Nintendo Wii Balance Platform: In addition to neurodevelopmental treatment, the cases are treated with virtual reality (VR) games on nintendo wii balance board for 8 weeks, 2 sessions a week. The VR games are performed twice in the first four weeks at the beginner level. During the following four weeks, advanced levels of the same games are selected and virtual reality therapy is performed with 2 repetitions.
  Interventions: Other: Exercise Interventions
- Hippotherapy Simulator Group: In addition to neurodevelopmental treatment, the cases are treated on a hippotherapy simulator for 8 weeks, 2 sessions a week. In the first 4 weeks, the warm-up and 1 speed intensities of the hippotherapy simulator are applied. During the next 4 weeks, cases are treated warm-up, 1, 2, 3, speed intensities, respectively.
  Interventions: Other: Exercise Interventions

INTERVENTIONS:
Other: Exercise Interventions — Rehabilitation methods and exercise practices to improve postural control in children with cerebral palsy. In addition to neurodevelopmental treatment, one group is treated with virtual reality games and the other group is treated with a hippotherapy simulator.

SUMMARY:
The aim of the research is to increase the active participation of children with Cerebral Palsy (CP) in therapy by integrating technological approaches into rehabilitation; To examine the effects of Nintendo Wii virtual reality games or hippotherapy simulator use on postural control, activity and participation in addition to Neurodevelopmental Therapy (NGT), which is frequently used in rehabilitation programs in CP, and to contribute to the relevant literature.

H1/H1-0: In the rehabilitation of children with Cerebral Palsy, Nintendo Wii virtual reality games in addition to NGT has or has no effect on postural control, lower extremity selective motor control, spasticity, activity and participation levels.

H2/H2-0: In the rehabilitation of children with Cerebral Palsy, Hippotherapy simulator in addition to NGT has or has no effect on postural control, lower extremity selective motor control, spasticity, activity and participation levels.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) defines a group of permanent disorders in the development of movement and posture, which occur in the developing fetal and newborn brain, due to non-progressive disorders, leading to activity limitations. The most common clinical type in CP is the spastic type, which is characterized by an increase in muscle tone. The deficiencies in the development of balance and protective reactions seen in children with spastic type CP, combined reactions and stereotypical movement patterns form the basis of postural control dysfunction. Postural control disorder results from primary brain injury that causes deficiencies in postural networks. motor networks; affected by spasticity, contracture, decreased force production, and abnormal timing; Perceptual networks are affected by deficiencies in the visual, tactile, proprioceptive, and vestibular systems. It is known to cause limitations during upper extremity activities, especially in gross motor skills that require balance such as walking.

Neurodevelopmental therapy (NGT); It is the most widely used method in CP rehabilitation all over the world, aiming to optimize function by improving postural control and facilitating the thought of movement. In a recent systematic review, the effects of treatment approaches in children with CP were examined and it was shown that technology-supported exercise training has a high level of evidence in improving gross motor functions. There are studies emphasizing that Nintendo Wii virtual reality games and hippotherapy simulator improve postural control and dynamic balance in children with CP.

Nintendo Wii virtual reality games and hippotherapy simulator are used as technology supported rehabilitation applications in addition to NGT in the research. Using both methods; In CP rehabilitation, the effects on the development of postural control, selective motor movement, spasticity level and, accordingly, activity and participation levels will be examined and contributed to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with spastic type CP,
* Being between the ages of 5-18,
* In Gross Motor Function Classification System (KMFSS); Taking place at I-II-III level,
* The family and the child agreed to participate in the study after reading the informed consent form.

Exclusion Criteria:

* Botulinum Toxin (BOTOX) injection to the lower extremity in the last 6 months,
* Having a diagnosis of epilepsy
* Having been diagnosed with mental retardation,
* Receiving additional treatment other than neurodevelopmental treatment,
* Having a vision and/or hearing problem that may affect participation in treatment methods.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between the ages of 5 and 18 who have been diagnosed with spastic cerebral palsy constitute the population of the study.
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Trunk Control Measurement Scale (TCMS) | Baseline and after 8 weeks
  The Trunk Control Measurement Scale is a clinical tool to measure trunk control in children with cerebral palsy. The TCMS evaluates of static and dynamic sitting balance.
  TCMS consists of 15 questions in total. A higher score on this scale represents better performance, with a TCMS total score ranging from 0 to 58.
  We will use this scale at the beginning and end of our study (after 8 weeks) so that we can see the effectiveness of the treatment methods we will apply.
Selective Control Assessment of the Lower Extremity (SCALE) | Baseline and after 8 weeks
  The Selective Control Assessment of the Lower Extremity (SCALE) is a clinical tool developed to quantify selective voluntary motor control (SVMC) in patients with cerebral palsy (CP). Hip, knee, ankle, subtalar, and toe joints are assessed bilaterally.
  We will use this scale at the beginning and end of our study (after 8 weeks) so that we can see the effectiveness of the treatment methods we will apply.
Modified Ashworth Scale (MAS) | Baseline and after 8 weeks
  The Modified Ashworth Scale is the most universally accepted clinical tool used to measure the increase of muscle tone. Hip flexors, hip adductors, knee flexors and ankle plantar flexor muscles in the lower extremities of the cases are evaluated bilaterally.
  We will use this scale at the beginning and end of our study (after 8 weeks) so that we can see the effectiveness of the treatment methods we will apply.
BeCure Balance Assessment System | Baseline and after 8 weeks
  The developed system evaluates the person's static standing balance, body center of gravity, load distributions in each foot, postural sway and proprioception. Evaluations made on the Nintendo Wii balance platform can be made as one foot-two feet, eyes open-closed, with or without images.
  We will use this scale at the beginning and end of our study (after 8 weeks) so that we can see the effectiveness of the treatment methods we will apply.

SECONDARY OUTCOMES:
Pediatric Evaluation of Disability Inventory (PEDI) | Baseline and after 8 weeks
  The Pediatric Evaluation of Disability Inventory (PEDI) is primarily designed for the functional evaluation of young children. Assessment is made by giving a score of '1' to the activities that the child can do, and '0' to the activities that the child cannot do, in the presence of the caregiver. It is seen that the total score increases with the increase in the functional independence level of the child.
  We will use this scale at the beginning and end of our study (after 8 weeks) so that we can see the effectiveness of the treatment methods we will apply.
Pediatric Quality of Life Inventory™ (PedsQL) 3.0 CP Module | Baseline and after 8 weeks
  PedsQL 3.0 CP Module is a scale developed to evaluate the quality of life domains of children with cerebral palsy between the ages of 2-18. The PedsQL 3.0 CP Module consists of seven subsections, a total of 35 items. Daily activities (9 items), school activities (4 items), movement and balance (5 items), pain and hurt (4 items), fatigue (4 items), eating activities (5 items) and speech and communication (4 items) ) consists of parts.
  We will use this scale at the beginning and end of our study (after 8 weeks) so that we can see the effectiveness of the treatment methods we will apply.

CONTACTS AND LOCATIONS:
Overall Officials: Yonca Zenginler Yazgan, Asst.Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No